CLINICAL TRIAL: NCT07006129
Title: Effectiveness of Perineorrhaphy in Pelvic Organ Prolapse Surgery
Acronym: PINPOPS
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: EPMDnr 2023-00177-01 (Study 1)
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Pelvic Organ Prolapse Vaginal Surgery; Pelvic Organ Prolapse (POP)
Keywords: Target Trial Emulation; Pelvic organ prolapse; Perineorrhaphy; Vaginal surgery; Cystocele; Rectocele; Apical prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse; Cystocele; Rectocele

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Perineorrhaphy: Primary pelvic organ prolapse surgery (no concomitant hysterectomy) with native tissue repair including perineorrhaphy
  Interventions: Procedure: Perineorrhaphy
- No perineorrhaphy: Primary pelvic organ prolapse surgery (no concomitant hysterectomy) with native tissue repair excluding perineorrhaphy
  Interventions: Procedure: No perineorrhaphy

INTERVENTIONS:
Procedure: Perineorrhaphy — Concomitant perineorrhaphy
  Groups: Perineorrhaphy
Procedure: No perineorrhaphy — No concomitant perineorrhaphy
  Groups: No perineorrhaphy

SUMMARY:
This is an observational registry-based study of long-term outcome after vaginal native tissue repair for pelvic organ prolapse designed to emulate a pragmatic open-label two-arm trial for which patients, in whom perineorrhaphy is not strictly indicated but clinically tenable, perioperatively are randomized to concomitant perineorrhaphy or not.

DETAILED DESCRIPTION:
This is an emulated pragmatic open-label two-arm trial in patients undergoing native tissue repair surgery for pelvic organ prolapse, in which patients are randomized perioperatively to either concomitant perineorrhaphy or not. The target population is the large group of patients for whom, at the discretion of the surgeon, this intervention is currently an option while not being strictly indicated. The investigators assumed that women were randomly assigned perioperatively to either strategy within levels of baseline co-variables: age, BMI, parity, lung disease, ASA-classification, constipation, hypermobility, prolapse in which vaginal compartment and if surgery is performed on it, year of primary surgery and region. Data was obtained from The Swedish National Quality Register of Gynaecological Surgery (GynOp), the Swedish National Patient Register, the Swedish Medical Birth Register, and the Swedish Cause of Death Register. In order to emulate a target trial, multiple imputation of missing data is followed by controlling for confounding through inverse probability weighting (IPW) in order to estimate the average treatment effect (ATE) in the primary analysis. In the secondary analysis, the primary analysis will be repeated but with overlap weights. Additional analyses: The sample will be re-weighted using IPW to estimate the average treatment effect on the treated (ATT). Restricted mean survival time (RMST) will be calculated at five years of follow-up for the primary outcome. Bias analysis: Mortality during follow up for the primary outcome will be used as a negative control.

ELIGIBILITY:
Inclusion Criteria:

* Pelvic organ prolapse surgery with vaginal native tissue repair without concomitant hysterectomy.

Exclusion Criteria:

* Primary surgery with colpocleisis, use of mesh, laparoscopic or abdominal surgery, concomitant incontinence surgery (eg transvaginal tape).
* Previous hysterectomy
* Previous pelvic organ prolapse surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with their primary vaginal pelvic organ prolapse surgery registered in the Swedish National Quality Register of Gynaecological Surgery (GynOp).
Sampling Method: Non-Probability Sample
Enrollment: 40646 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Reoperation | 5 years
  Reported as absolute risk difference, with cumulative risks during five years of follow-up estimated using the Kaplan-Meier estimator.
  Data obtained from the The Swedish National Quality Register of Gynaecological Surgery (GynOp) and the Swedish National Patient Register.

SECONDARY OUTCOMES:
Symptoms of a vaginal bulge (patient reported outcome) | At 1 year
  Absolute risk difference for the outcome at 1 year follow-up with the non-inferiority margin set to 10% of the absolute risk in the comparison group. Data obtained from the The Swedish National Quality Register of Gynaecological Surgery (GynOp).
Unsatisfied (patient reported outcome) | At 1 year
  Absolute risk difference for the outcome at 1 year follow-up with the non-inferiority margin set to 10% of the absolute risk in the comparison group. Data obtained from the The Swedish National Quality Register of Gynaecological Surgery (GynOp).

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No
Data are available from the registry source.